CLINICAL TRIAL: NCT04579731
Title: Development of Fecal Scoring for the Management of Fecal Impaction With Regards to Lower Urinary Tract Dysfunction
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kwanjin Park, Associate Professor, Seoul National University Hospital
Other Study IDs: 2008-133-1150
Record Dates: First submitted 2020-09-21; First posted 2020-10-08 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Fecal Impaction; Lower Urinary Tract Disorder; Bladder Dysfunction; Bowel Dysfunction
MeSH Terms: conditions — Fecal Impaction; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fecal Impaction (LUTD-FI): Patients with both significant Lower Urinary Tract Dysfunction history suggestive of constipation were treated with lactitol monohydrate syrup 10 g for eight weeks. Following eight weeks of treatment, patients were re-evaluated and those with 50% of symptom improvement were assumed to have a significant improvement attributable to the development of Lower Urinary Tract Dysfunction- Fecal Impaction (LUTD-FI).
- Lower Urinary Tract Dysfunction Not Related to Fecal Impaction: Patients with both significant Lower Urinary Tract Dysfunction history suggestive of constipation were treated with lactitol monohydrate syrup 10 g for eight weeks. Following eight weeks of treatment, patients were re-evaluated and those without symptom improvement place into lower urinary tract dysfunction not related to fecal impaction (LUTD-FI). They serve as a control group.
  Interventions: Drug: Lactitol Monohydrate

INTERVENTIONS:
Drug: Lactitol Monohydrate — Patients with lower urinary tract dysfunction and assumed to have constipation were placed on lactitol monohydrate 10 g for 8 weeks, and had re-evaluated.
  Groups: Lower Urinary Tract Dysfunction Not Related to Fecal Impaction

SUMMARY:
The role of bowel bladder disorder, or BBD, has been highlighted as a major player in vesicoureteral reflux and urinary tract infection (UTI). However, the diagnosis of BBD are still conceptual and subjective, because of the diagnosis of constipation, main pathophysiology in BBD has not been established well.

DETAILED DESCRIPTION:
Functional constipation is a common disorder among children, accounting for 3-5% of visits to pediatric clinics and even 10% to 25% of consultation for pediatric gastroenterologists. It could cause recurrent abdominal pain, stool retention as well as fecal incontinence. In the urologic field, this is known to develop urinary symptoms. Constipation has been associated with voiding dysfunction and urinary tract infection in children. It is assumed that impacted stool in distal rectum mechanically affect the bladder leading to detrusor overactivity. Additionally, impacted stool would elevate the uretheral sphincter tone, having patients void with incomplete sphincter relaxation and eliciting dysfunctional voiding. Stool impaction may be the source of bacteria causing urinary tract infection and led to recurrent bacteriuria. Treatment of constipation by itself is quite effective alleviating urologic symptoms in as much as two-third of the patients.

The role of constipation has been highlighted as a major player in vesicoureteral reflux and urinary tract infection (UTI). The presence of bowel bladder disorder (BBD) was associated with higher risk of breakthrough infection and a lack of spontaneous resolution. Although constipation is the major player in BBC, there is any objective standard regarding the diagnosis and treatment of constipation. Given the high prevalence and morbidity of children affected by UTI or VUR in relations to BBD, it is imperative that diagnostic and treatment methods are developed.

Despite the known implication of constipation, the diagnosis of constipation may be problematic due to a lack of standard definition for this condition. This may be due to different views between clinicians about which aspect are most crucial for diagnosing constipation. Some underline the subjective nature such as infrequent or difficult defecation, other stress the quality of stool, still others were in search of objective criteria of constipation, like the amount of impacted stool or colonic transit time. Consequently, various criteria have been reported.

The lack of standard criteria for constipation causes trouble sometimes in making a proper decision for diagnosis, intervention, follow-up, and discharge of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with having both significant Lowery Urinary Tract Dysfunction history suggestive of constipation (more than two positive criteria in ROME 4).
* Parental recalling of hard stool (Bristol stool scale of 6 or 7).
* Parental impression of constipation.

Exclusion Criteria:

- Those without Lower Urinary Tract Dysfunction or constipation.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who visited the department of pediatric urology for significant lower urinary tract dysfunction with history suggestive of constipation.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
KUB (Kidneys, Ureters, Bladder) | After 8 weeks from the baseline
  Examine the outcomes of the treatment of lactitol monohydrate 10 g in relation to Lower Urinary Tract Dysfunction and fecal impaction by using KUB (Kidneys, Ureters, Bladder) x-ray images.

CONTACTS AND LOCATIONS:
Overall Officials: Kwanjin Park, M.D. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No